CLINICAL TRIAL: NCT01503307
Title: Parenting After Infant Congenital Heart Defect Diagnosis
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Children's Hospital and Health System Foundation, Wisconsin (Other); University of Wisconsin, Madison (Other); University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: CHW 08/160; GC 728 (Other: Medical College of Wisconsin)
Record Dates: First submitted 2011-12-28; First posted 2012-01-04 (Estimated); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Congenital Heart Disease
Keywords: prenatal chd diagnosis; postpartum chd diagnosis; parenting; internal working models
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Prenatal/Postpartum CHD Diagnosis: parent of a baby (prenatal or postpartum)who was recently found to have a heart defect.

SUMMARY:
The purpose of this research study is to learn about parents' experiences following diagnosis of a fetal/neonatal Congenital Heart Defect (CHD). Nurses, physicians, and other health-care clinicians will benefit from an improved understanding of what the diagnosis means to parents and what they expect concerning the infant, being a parent, and caregiving tasks and responsibilities. The investigators expect that the knowledge gained will increase clinicians' ability to respond to parents' needs.

DETAILED DESCRIPTION:
Parental mental health status is linked to the development and quality of caregiving, as well as physiological and psychosocial outcomes for the infant/child with a heart defect.

This is an evolving population of parents with most challenged prenatally with a fetal diagnosis and later as caregivers for medically complex infants. Parents with pre- and postnatally diagnosed infants are at risk for sub-optimal mental health. Parents' experiences and needs differ by timing of diagnosis.

Several gaps in the literature exist. First, advances in technology raise questions about how becoming a caregiver is experienced considering the timing of the diagnosis. Second, little is known about how the timing of the diagnosis could influence parents' mental health status and caregiving after diagnosis. Finally, more study is needed to identify the type, timing and duration of intervention to support these parents as caregivers and optimize their infants' health.

Data collected for this study included demographic and health information (from parents and infant health records), measures of distress (symptoms of depression, anxiety and trauma), and interviews. Semi-structured interviews were conducted with parents in person in the hospital and home settings. Interviews with each couple in the prenatally diagnosed group were conducted once during the third trimester of pregnancy and once within 12 weeks after birth. Interviews with each couple or mother in the postnatally diagnosed group were conducted once within 12 weeks after birth. Interviews lasted 1-3 hours, were audio-recorded and transcribed verbatim for analysis. Field notes were also written and audio recorded for use in analysis.

Directed content analysis has been used to describe parents' experiences and caregiving motivations in relation to parental distress and severity of infant illness. Analysis of data is ongoing. Additional analyses are expected to further improve knowledge on the differing needs of parents of pre- and postnatally diagnosed infants, as well as parents' experiences and caregiving motivations in the context of discharge from tertiary care.

ELIGIBILITY:
Inclusion Criteria for Parents:

* at least 18 years old
* English speaking and reading
* not known to have a mental illness or cognitive deficit

Inclusion Criteria for Infant:

* prenatal or postnatal diagnosis of a complex CHD that requires surgical repair or palliation early in the infant's life (i.e., tetralogy of Fallot, atrial-ventricular canal, ventricular septal defect, pulmonary stenosis, tricuspid atresia, hypoplastic right or left heart, or other complex condition). Infants will not be excluded if they also have congenital syndromes or extra-cardiac defects.

Exclusion Criteria:

* no CHD diagnosis

Max Age: 12 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: In this year-long study, 12 to 16 families (mothers and fathers) will be recruited-6 to 8 of the families from the fetal diagnosis clinic at either Meriter Hospital or Children's Hospital of Wisconsin and 6 to 8 families whose infant is diagnosed soon after birth with a complex CHD at either Meriter Hospital or Children's Hospital of Wisconsin.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Creation of a typology of perinatal internal working models of parenting in congenital heart disease. | 1 year
  Qualitative analysis of interviews.

SECONDARY OUTCOMES:
Parent outcomes | 1 year
  Impact of Event Scale - Stress Reactions Center for Epidemiologic Studies Depression Scale - Depression State-Trait Anxiety Inventory - Anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Karen Pridham, PhD, RN, Principal Investigator — University of Wisconsin, Madison; Anne C McKechnie, PhD, RN, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - University of Wisconsin Madison, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin